CLINICAL TRIAL: NCT05946772
Title: Cyclosporine In Takotsubo Syndrome (CIT) Trial
Brief Title: Cyclosporine In Takotsubo Syndrome
Acronym: CIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Centre of Cardiovascular Research (DZHK) (Unknown); Coordinating Centre for Clinical Studies (KKS) Heidelberg (Unknown)
Responsible Party: Principal Investigator, Norbert Frey, MD, Professor Dr. Norbert Frey, MD, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DZHK29; DZHK29 (Other Grant/Funding Number: German Centre of Cardiovascular Research (DZHK))
Record Dates: First submitted 2023-06-19; First posted 2023-07-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: Takotsubo syndrome; Troponin; Cyclosporine; Inflammation; Acute heart failure
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Inflammation | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: Double-blind multicentre RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, care providers, and outcomes assessors are masked from study arm affiliation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): A concealed 0.9% sodium chloride (NaCl) preparation will be applied intravenously at baseline, 12h, and 24h.
  Interventions: Drug: Placebo
- CsA (Experimental): Cyclosporine A will be applied intravenously at baseline, 12h, and 24h.
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: Cyclosporine A — 2.5mg/kg body weight Cyclosporine A as an intravenous bolus
  Arms: CsA
Drug: Placebo — The same amount of 0.9% sodium chloride (NaCl0.9%) will be applied in an indistinguishable package as an intravenous bolus
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the impact of repetitive acute Cyclosporine A (CsA) bolus therapy in patients suffering from TTS with an elevated risk of impaired outcome. The main question it aims to answer is whether CsA reduces myocardial injury (primary outcome). Participants will receive CsA or placebo at baseline and every 12h in the first 24h after study inclusion. Researchers will compare CsA and the placebo group to see if a) myocardial injury is reduced, and b) ejection fraction is improved compared to baseline, as well as several other secondary endpoints over a one year follow-up.

DETAILED DESCRIPTION:
Takotsubo syndrome (TTS) has been suggested to be caused by catecholamine excess with myocardial inflammation-enhanced cardiac injury. Substantial morbidity and mortality have repeatedly been reported, even though reduced ejection fraction frequently recovers spontaneously. So far there is no evidence-based treatment available. In a clinically relevant mouse model of catecholamine-driven TTS, cyclosporine A (CsA) bolus therapy markedly improves outcome, likely mediated via suppression of calcineurin-driven inflammation. The investigators have thus designed a pilot multicentre randomized controlled trial (RCT) to investigate the impact of repetitive CsA bolus therapy vs. placebo in acute TTS patients with an increased risk of intrahospital complications and a 32% estimated 5-year mortality. As primary outcome myocardial damage will be compared between groups via high-sensitive Troponin T plasma area under the curve (AUC). Recovery of cardiac function, the extent of myocardial oedema at 72h, length of hospital-stay, 30-day-, and 1-year composite clinical outcome as well as psychosocial and quality of life self-assessment will be secondary endpoints. The results of this trial may reveal CsA as a first pathophysiology-driven treatment option of TTS and enable a phase III follow-up trial with outcome parameters as primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years)
2. Symptom onset < 24h
3. With a high probability of TTS:

   1. InterTAK Diagnostic Score > 39 and
   2. Regional wall motion abnormality (WMA) consistent with TTS; no coronary intervention (PCI), or reperfused myocardial ischemia according to MRI
4. With a high probability of impaired outcome:

   1. InterTAK Prognostic Score >15 or
   2. GEIST Score > 19

Exclusion Criteria:

1. Suspected infection
2. Cardiac arrest, ventricular fibrillation, invasive ventilatory support
3. Known hypersensitivity to CsA, egg, peanut, or soya-bean proteins
4. Renal insufficiency (creatinin clearance < 30 ml/min/1.73m²)
5. Liver insufficiency
6. Uncontrolled hypertension (>180/110 mmHg)
7. Hypericum perforatum, Stiripentol, Aliskiren, Bosentan, or Rosuvastatin treatment
8. Pregnancy or women of childbearing age without contraception
9. Any disorder associated with immunological dysfunction < 6 months prior to presentation
10. Immunosuppressive therapy
11. Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Myocardial damage | baseline, hour 3, hour 12, hour 24, hour 36, hour 48, hour 60, hour 72, day 30
  High-sensitive Troponin T AUC over several time points between CsA and Placebo.

SECONDARY OUTCOMES:
Change in Ejection fraction from baseline | baseline, hour 24, hour 48, hour 72, day 30
  Multiple timepoints will be compared to baseline between CsA and Placebo.
Fold-change in Troponin plasma concentration | baseline, hour 3, hour 12, hour 24, hour 36, hour 48, hour 60, hour 72, day 30
  The change of high-sensitive Troponin T will be compared to baseline between CsA and Placebo for multiple time points.
Fold-change in creatine kinase plasma concentration | baseline, hour 3, hour 12, hour 24, hour 36, hour 48, hour 60, hour 72, day 30
  The change of creatine kinase will be compared to baseline between CsA and Placebo for multiple time points.
Fold-change in NTproBNP plasma concentration | baseline, hour 3, hour 12, hour 24, hour 36, hour 48, hour 60, hour 72, day 30
  The change of NTproBNP will be compared to baseline between CsA and Placebo for multiple time points.
Fold-change in interleukin-6 plasma concentration | baseline, hour 12, hour 24, hour 36, hour 48, hour 60, hour 72, day 30
  The change of interleukin-6 will be compared to baseline between CsA and Placebo for multiple time points.
Fold-change in procalcitonin plasma concentration | baseline, hour 12, hour 24, hour 36, hour 48, hour 60, hour 72, day 30
  The change of procalcitonin will be compared to baseline between CsA and Placebo for multiple time points.
Myocardial edema | hour 72
  Cardiac MRI will be used to assess the T2 signal intensity ratio for comparison between CsA and Placebo at 72h.
Myocardial inflammation | hour 72
  Cardiac MRI will be used to assess the early gadolinium enhancement ratio for comparison between CsA and Placebo at 72h.
Rate of cardiovascular events at day 30 | day 30
  At day 30 a composite cardiovascular outcome measure includes overall mortality, stroke, myocardial infarction, heart failure hospitalization, recurrent TTS, cardiac arrest, ventricular fibrillation, ventricular tachycardia, novel atrial fibrillation, and thromboembolism. The measure is considered positive if one of the above occurs. The amount of patients with positive and negative events is then compared between the CsA and placebo arm.
Rate of cardiovascular events at 1 year | 1 year
  At 1 year a composite cardiovascular outcome measure includes overall mortality, stroke, myocardial infarction, heart failure hospitalization, recurrent TTS, cardiac arrest, ventricular fibrillation, ventricular tachycardia, novel atrial fibrillation, and thromboembolism. The measure is considered positive if one of the above occurs. The amount of patients with positive and negative events is then compared between the CsA and placebo arm.
Rate of novel disease onset | day 30 and at 1 year
  At 30 days and 1-year novel clinical diagnoses during follow-up including cancer or neurological diseases will be assessed.
Symptom burden at day 30 | day 30
  Patient-reported outcome will be quantified by the Kansas City Cardiomyopathy Questionnaire after 30d and 1 year (scale 0-100 points: 0-24 points: very poor; 25-49 points: poor; 50-74 points: fair; 75-100: good).
Symptom burden at 1 year | 1 year
  Patient-reported outcome will be quantified by the Kansas City Cardiomyopathy Questionnaire at 1 year (scale 0-100 points: 0-24 points: very poor; 25-49 points: poor; 50-74 points: fair; 75-100: good).
Depression score at day 30 | day 30
  Patient-reported psychosocial assessment will be quantified by the well validated German patient health questionnaire 9 (PHQ-9) scale (range 0-27 points, higher points indicate worse depressive symptoms).
Depression score at year 1 | 1 year
  Patient-reported psychosocial assessment will be quantified by the well validated German patient health questionnaire 9 (PHQ-9) scale (range 0-27 points, higher points indicate worse depressive symptoms).
Anxiety score at day 30 | day 30
  Patient-reported psychosocial assessment will be quantified by the well validated German generalized anxiety disorder 7 (GAD-7) questionnaire (range 0-21 points, higher points indicate worse anxiety).
Anxiety score at year 1 | year 1
  Patient-reported psychosocial assessment will be quantified by the well validated German generalized anxiety disorder 7 (GAD-7) questionnaire (range 0-21 points, higher points indicate worse anxiety).
PTSD score at 30 days | day 30
  Patient-reported psychosocial assessment will be quantified by the well validated German primary care posttraumatic stress disorder questionnaire 5 (PC-PTSD-5) (0-5 points, higher points indicate more symptoms of posttraumatic stress disorder).
PTSD score at 1 year | year 1
  Patient-reported psychosocial assessment will be quantified by the well validated German primary care posttraumatic stress disorder questionnaire 5 (PC-PTSD-5) (0-5 points, higher points indicate more symptoms of posttraumatic stress disorder).
Length of intermediate care or intensive care unit stay | day 30
  Length of intermediate care or intensive care unit stay will be compared between groups
Length of hospital stay | day 30
  Length of hospital stay will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Frey, MD, Principal Investigator — University Hospital Heidelberg; Bastian Bruns, MD, Principal Investigator — University Hospital Heidelberg
Locations (21):
- Germany (21):
  - Kerckhoff Heart Center, Bad Nauheim / Gießen University, Bad Nauheim
  - Department of Cardiology, Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Department of Cardiology, Charité - Universitätsmedizin Berlin, Berlin
  - Heart Centre - University Hospital Bonn, Bonn
  - Department of Cardiology, University Hospital Köln, Cologne
  - Department of Cardiology, University Hospital Dresden, Dresden
  - Cardiovascular Centre - University Hospital Düsseldorf, Düsseldorf
  - Department of Cardiology - University Hospital Essen, Essen
  - University Medical Center Göttingen, Göttingen
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Department of Cardiology, University Hospital Hannover, Hanover
  - Department of Cardiology, Heidelberg University Hospital, Heidelberg
  - University Medical Center Schleswig-Holstein/Campus Kiel, Kiel
  - Leipzig Heart Center, Leipzig
  - University Medical Center Schleswig-Holstein/Campus Lübeck, Lübeck
  - Department of Cardiology, University Hospital Magdeburg, Magdeburg
  - Department of Cardiology, University Hospital Mainz, Mainz
  - Department of Cardiology, University Hospital Mannheim, Mannheim
  - Department of Cardiology, Hospital of the Ludwig-Maximilians-University Munich, München
  - University Hospital rechts der Isar, Technical University of Munich, München
  - Department of Cardiology, University Hospital Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruns B, Elsous N, Burghaus I, Steyrer K, Joos M, Kramer T, Scheffel M, Blankenberg S, Eitel I, Massberg S, Thiele H, Meder B, Backs J, Frey N. Rationale and design of the cyclosporine in Takotsubo syndrome (CIT) trial. Am Heart J. 2025 Nov;289:147-157. doi: 10.1016/j.ahj.2025.04.020. Epub 2025 Apr 21. PMID 40268179